CLINICAL TRIAL: NCT00788593
Title: A Randomized, Double-Blind, Dose Response-Control, Crossover Study to Evaluate the Safety and Efficacy of Two Doses of EUR-1008 in Chronic Pancreatitis (CP) Patients With Exocrine Pancreatic Insufficiency (EPI)
Brief Title: A Randomized, Double-Blind, Dose Response-Control, Crossover Study to Evaluate the Safety and Efficacy of Two Doses of EUR-1008 (APT-1008) in Chronic Pancreatitis (CP) Participants With Exocrine Pancreatic Insufficiency (EPI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-002
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Pancreatitis; Exocrine Pancreatic Insufficiency
Keywords: Chronic Pancreatitis; Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- EUR-1008 (APT-1008) High Dose (Experimental)
  Interventions: Drug: EUR-1008 (APT-1008) High Dose
- EUR-1008 (APT-1008) Low Dose (Experimental)
  Interventions: Drug: EUR-1008 (APT-1008) Low Dose

INTERVENTIONS:
Drug: Placebo — Placebo matching to EUR-1008 (APT-1008) capsules orally daily for 4 days home treatment and 3 to 5 days hospital treatment in the baseline run-in phase, which will then be randomized to either high dose or low dose of EUR-1008 (APT-1008).
  Arms: Placebo
Drug: EUR-1008 (APT-1008) High Dose — EUR-1008 (APT-1008) total high dose 140,000 lipase USP Lipase units will be given as 7 capsules containing 20,000 USP Lipase units each, orally daily, distributed over the day per gram of fat in diet (possible example: 2 capsules with breakfast, 2 capsules with lunch, 2 capsules with dinner and 1 capsule with a snack) for 6 days home treatment and 3 to 5 days hospital treatment in either first intervention period or second intervention period.
  Other Names: Zenpep
  Arms: EUR-1008 (APT-1008) High Dose
Drug: EUR-1008 (APT-1008) Low Dose — EUR-1008 (APT-1008) total low dose 35,000 lipase USP Lipase units will be given as 7 capsules containing 5,000 USP Lipase units each, orally daily, distributed over the day per gram of fat in diet (possible example: 2 capsules with breakfast, 2 capsules with lunch, 2 capsules with dinner and 1 capsule with a snack) for 6 days home treatment and 3 to 5 days hospital treatment in either first intervention period or second intervention period.
  Other Names: Zenpep
  Arms: EUR-1008 (APT-1008) Low Dose

SUMMARY:
The primary efficacy objective of this study is to evaluate the difference in coefficient of fat absorption (CFA) of participants treated with high dose EUR-1008 (APT-1008) versus low dose of EUR-1008 (APT-1008) in the treatment of signs and symptoms of malabsorption in participants with EPI associated with CP. This study is sponsored by Aptalis Pharma (formerly Eurand).

DETAILED DESCRIPTION:
After screening, eligible participants will start the placebo baseline ambulatory phase (4 days). On day 5, they will be hospitalized for three to five days, to undergo a "baseline" 72-hour CFA determination under a controlled diet and using a stool marker to indicate the beginning and end of the controlled diet period, while they continue receiving placebo treatment. At the end of the placebo baseline phase, participants will be randomized to a "high dose followed by a low dose" or to a "low dose followed by a high dose" EUR-1008 (APT-1008) dose sequence and proceed to the first crossover (treatment) phase. Each crossover (treatment) phase will consist of a stabilization period for six days at home, followed by a hospitalization of three to five days to undergo a 72-hour CFA determination using a controlled diet and using a stool marker to indicate the beginning and end of the controlled diet period.

Participants will immediately proceed from the first crossover (treatment) phase to the second without a washout period or return-to-baseline period in between phases. Participants will be stabilized at home for 6 days. Any residual lipase from the prior treatment phase is likely to be a negligible influence on the subsequent CFA determination because participants will be taking the new dose level (high or low) for six days before the beginning of sample collection for a new CFA. This interval is more than enough time for the CFA to be reflective of only the new dose.

ELIGIBILITY:
Inclusion Criteria:

* Participants are male or female
* Participants with age over 18 years
* Participants who have written, legally valid informed consent
* Women of childbearing potential must be using a medically acceptable form of birth control for the 30 days prior to the beginning of the study and agree to maintain adequate birth control measures during the whole duration of the study plus an additional 30 days as well as have a negative pregnancy test at screening Visit 3 and Visit 7
* Participants with documented diagnosis of CP by medical history and it is preferred that it is supported by imaging evidence confirming CP which include: abnormal endoscopic retrograde cholangio-pancreatography (ERCP) (Cambridge Class 4), abnormal computed tomography (CT) scan (dilated main pancreatic duct, atrophy of the pancreas or calcification), abnormal ultrasound, or endoscopic ultrasound with at least 5 abnormalities noted
* In the case of pancreatic surgery, the participant can be included with partial or distal resection of the pancreas (not due to cancer)
* Participants with documented EPI with target fecal elastase (FE) less than or equal to 100 microgram per gram (mcg/g) of stool using the monoclonal test (pancreatic elastase 1 [PE1] by Genova Diagnostics) performed at the screening visit. The mean coefficient of variation (CV) for the FE test is 20 percent (%)

Exclusion Criteria:

* Participants known to the investigator to have a significant medical and/or mental disease that would compromise the participant's welfare, pose an unacceptable risk to him/her or confound the study results
* Participants who participated in a clinical trial within 30 days of randomization or per specific country regulations/guidelines
* Participants with cystic fibrosis
* Participants with excessive alcohol consumption
* Participants with drug abuse
* Participants with contraindicated medications or who are unable to discontinue prohibited concomitant medication
* Participants with uncontrolled diabetes mellitus
* Participants allergic to pork protein/unwilling to ingest pork products
* Participants with atopic predisposition such as multiple drug hypersensitivity, allergic asthma, urticaria, or other relevant allergic diathesis
* Participants who are pregnant or lactating
* Participants with acute pancreatitis or acute exacerbation in chronic pancreatitis
* Participants with acute biliary disease
* Participants with malabsorption syndrome caused by a metabolic disease or by surgery, not related to exocrine pancreatic insufficiency
* Participants with any resection of the stomach or the gastrointestinal tract that will affect transit time and/or gastric emptying.
* Participants with evidence of active gastric or duodenal ulcer
* Participants with chronic inflammatory bowel disease
* Participants with any history of pancreatic cancer and other non-cutaneous malignancies (except basal cell and squamous cell carcinoma of the skin in situ that have been removed and not reoccurred in 5 years)
* Participants with viral hepatitis with infectious virions in blood and/or body fluids (any etiology)
* Participants with human immunodeficiency virus (HIV) infection
* Participants with hyperuricemia ( greater than [>] 1.5 times upper normal value for lab)
* Participants with any acute or chronic disease, which in the opinion of the investigator could influence study results or pose a risk to the participants' safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (18):
- United States (9):
  - Woodland International Research Group, Little Rock, Arkansas
  - HealthCare Partners Medical Group, Los Angeles, California
  - University of Florida, General Clinical Research Center, Gainesville, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Veterans Affairs Edward Jr. Hines Hospital, Building #1, Hines, Illinois
  - University of Iowa Hospitals and Clinics, Iowa Ctiy, Iowa
  - University of Kentucky, Medical Center, Department of Gastroenterology, Lexington, Kentucky
  - University of Louisville, Carmichael Building, Louisville, Kentucky
  - University of Missouri Health Care, Columbia, Missouri
- Italy (4):
  - Dipartmento di Malattie dell' apparato digerente e Medicina Interna- Unita Operativa di MedicinaInterna Corinaldesi Azienda Ospedaliero- Universitaria Policlinico Sant'Orsola Malpighi Via Massarenti, Massarenti, Bologna
  - Istituto Clinico Humanitas - Universita' Di Milano Via Manzoni, Rozzano, Milano
  - Istituto di Clinica Chirurgica (Ensoscopia Digestive Chirurgica) Policlinico Gemelli-Universita Cattolica del Sacro Cuore, Largo Agostino Gemelli, Roma
  - Centro Richerche Cliniche di Verona, Le Ludovico Scuro, Verona
- Ukraine (5):
  - Department of Therapy and Family Medicine of the Facility of Post graduate Education of Crimea State Medical University named after S.I. Georglyevskyy Republic Clinical Hospital named after M.O. Semashko, Simferopol, Autonomous Republic of Crimea
  - Department of Internal Medicine No 2 of Donetsk State University named after M. Gorkly, City Clinical Hospital No 3, Donetsk, Donetsk Oblast
  - Department of Liver and Gastrointestinal Tract Disease Institute of Therapy named after L.T. Maylaya of Academy of Medical Sciences of the Ukraine, Kharkiv, Kharklv
  - Department of Faculty Therapy No 1 with the Course of Postgraduate Training of Physicians for Gastroenterology and Endoscopy, National Medical University named after O.O. Bogomolets, City Hospital No 18, Kyiv, Kylv
  - General Therapy Clinic, Military Clinical Hospital of Ministry of Defense of Ukraine 18, Kyiv, Kylv

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Baseline: Placebo matched to EUR-1008 (APT-1008) capsules orally daily for 4 days home treatment and 3 to 5 days hospital treatment in the baseline run-in phase, which were then randomized to either high dose or low dose of EUR-1008 (APT-1008).
- EUR-1008 (APT-1008) High Dose, Then Low Dose: EUR-1008 (APT-1008) total high dose 140,000 lipase United States Pharmacopeia (USP) Lipase units was given as 7 capsules containing 20,000 USP Lipase units each, orally daily, as high dose in first intervention period followed by EUR-1008 (APT-1008) total low dose 35,000 lipase USP Lipase units was given as 7 capsules containing 5,000 USP Lipase units each, orally daily, as low dose in second intervention period; 7 capsules were distributed over the day per gram of fat in diet (possible example: 2 capsules with breakfast, 2 capsules with lunch, 2 capsules with dinner and 1 capsule with a snack) for 6 days home treatment and 3 to 5 days hospital treatment.
- EUR-1008 (APT-1008) Low Dose, Then High Dose: EUR-1008 (APT-1008) total low dose 35,000 lipase USP Lipase units was given as 7 capsules containing 5,000 USP Lipase units each, orally daily, as high dose in first intervention period followed by EUR-1008 (APT-1008) total high dose 140,000 lipase United States Pharmacopeia (USP) Lipase units was given as 7 capsules containing 20,000 USP Lipase units each, orally daily, as low dose in second intervention period; 7 capsules were distributed over the day per gram of fat in diet (possible example: 2 capsules with breakfast, 2 capsules with lunch, 2 capsules with dinner and 1 capsule with a snack) for 6 days home treatment and 3 to 5 days hospital treatment.
Period: Placebo Run-in Phase
Arm/Group | Placebo Baseline | EUR-1008 (APT-1008) High Dose, Then Low Dose | EUR-1008 (APT-1008) Low Dose, Then High Dose
Started | 82 | 0 | 0
Completed | 76 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Period: First Intervention Period
Arm/Group | Placebo Baseline | EUR-1008 (APT-1008) High Dose, Then Low Dose | EUR-1008 (APT-1008) Low Dose, Then High Dose
Started | 0 | 39 | 37
Completed | 0 | 38 | 37
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Second Intervention Period
Arm/Group | Placebo Baseline | EUR-1008 (APT-1008) High Dose, Then Low Dose | EUR-1008 (APT-1008) Low Dose, Then High Dose
Started | 0 | 38 | 37
Completed | 0 | 37 | 36
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least 1 dose of the study medication.
Groups:
- Entire Study Population: Includes participants who received placebo, EUR-1008 (APT-1008) high dose first and EUR-1008 (APT-1008) low dose first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.91 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 53
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 68.75 (14.12)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2).
  kg/m^2 | 23.36 (4.44)

OUTCOME MEASURES:

1. Primary Outcome: Percent Coefficient of Fat Absorption (CFA) of Participants Treated With High Dose EUR-1008 and Low Dose EUR-1008
Description: Percent CFA was calculated as ([fat intake - fat excretion]/fat intake)*100, determined in the stools collected during the 72-hour CFA determination period. Mean percent CFA was calculated for the 3 to 5 days of hospital treatment in first and second intervention periods.
Time Frame: 3 to 5 days of hospital treatment in first and second intervention periods
Population: FAS included all participants who received at least 1 dose of the study medication. Here "N" (number of participants analyzed) signifies those participants for whom the CFA values were available.
Measure: Mean (Standard Deviation); unit: percent CFA
Groups:
- EUR-1008 (APT-1008) Low Dose: EUR-1008 (APT-1008) total low dose 35,000 lipase USP Lipase units was given as 7 capsules containing 5,000 USP Lipase units each, orally daily, distributed over the day per gram of fat in diet (possible example: 2 capsules with breakfast, 2 capsules with lunch, 2 capsules with dinner and 1 capsule with a snack) for 6 days home treatment and 3 to 5 days hospital treatment in either first intervention period or second intervention period.
- EUR-1008 (APT-1008) High Dose: EUR-1008 (APT-1008) total high dose 140,000 lipase USP Lipase units was given as 7 capsules containing 20,000 USP Lipase units each, orally daily, distributed over the day per gram of fat in diet (possible example: 2 capsules with breakfast, 2 capsules with lunch, 2 capsules with dinner and 1 capsule with a snack) for 6 days home treatment and 3 to 5 days hospital treatment in either first intervention period or second intervention period.
Arm/Group | EUR-1008 (APT-1008) Low Dose | EUR-1008 (APT-1008) High Dose
Number analyzed (Participants) | 72 | 72
percent CFA | 88.87 (12.44) | 89.86 (8.77) [-0.656 to 2.701]
Statistical Analysis 1: Comparison: EUR-1008 (APT-1008) Low Dose vs EUR-1008 (APT-1008) High Dose; Treatment difference and 95 percent (%) confidence interval (CI) was based on LS mean from analysis of covariance (ANCOVA) which included participant as random effect, treatment, period and sequence as fixed effects, and placebo baseline CFA value as covariate; Test type: Superiority or Other; p = 0.228, ANCOVA; Least Square (LS) Mean Difference = 1.023, 95% CI 2-sided [-0.656 to 2.701]

2. Secondary Outcome: Change From Placebo Baseline in Percent Coefficient of Fat Absorption (CFA) in High Dose EUR-1008 and Low Dose EUR-1008 During Hospital Treatment
Description: Percent CFA was calculated as ([fat intake - fat excretion]/fat intake)*100, determined in the stools collected during the 72-hour CFA determination period. Mean percent CFA was calculated for 3 to 5 days of hospital treatment in first and second intervention periods.
Time Frame: Baseline, 3 to 5 days of hospital treatment in first and second intervention periods
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent CFA
Groups:
- Placebo Baseline: Placebo matched to EUR-1008 (APT-1008) capsules, orally daily, for 4 days home treatment and 3 to 5 days hospital treatment in the baseline run-in phase, which were then randomized to either high dose or low dose of EUR-1008 (APT-1008)
Arm/Group | Placebo Baseline | EUR-1008 (APT-1008) Low Dose | EUR-1008 (APT-1008) High Dose
Number analyzed (Participants) | 82 | 72 | 72
percent CFA
  Baseline | 81.68 (22.13) | NA (NA) — Data was not reported as EUR-1008 low dose was not given at baseline. | NA (NA) — Data was not reported as EUR-1008 high dose was not given at baseline.
  Change During Hospital Period | NA (NA) — Data was not reported as placebo was not given during hospital treatment period. | 7.19 (14.49) | 8.18 (17.35)
Statistical Analysis 1: Comparison: Placebo Baseline vs EUR-1008 (APT-1008) Low Dose; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo Baseline vs EUR-1008 (APT-1008) High Dose; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change From Placebo Baseline in Percent Coefficient of Nitrogen Absorption (CNA) During Hospital Treatment
Description: Percent CNA was calculated as [(nitrogen intake - nitrogen excretion)/nitrogen intake]*100 , determined in the stools collected during the 72-hour CNA determination period. Nitrogen intake was calculated as protein intake/6.2. Nitrogen excretion was measured as total fecal nitrogen. Mean percent CNA was calculated for 3 to 5 days of hospital treatment in first and second intervention periods.
Time Frame: Baseline, 3 to 5 days of hospital treatment in first and second intervention periods
Population: FAS included all participants who received at least one dose of the study drug. Here "N" (number of participants analyzed) represents number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent CNA
Arm/Group | Placebo Baseline | EUR-1008 (APT-1008) Low Dose | EUR-1008 (APT-1008) High Dose
Number analyzed (Participants) | 82 | 74 | 75
percent CNA
  Baseline | 78.05 (18.64) | NA (NA) — Data was not reported as EUR-1008 low dose was not given at baseline. | NA (NA) — Data was not reported as EUR-1008 high dose was not given at baseline.
  Change During Hospital Period | NA (NA) — Data was not reported as placebo was not given during hospital treatment period. | 5.33 (10.38) | 7.62 (15.55)
Statistical Analysis 1: Comparison: Placebo Baseline vs EUR-1008 (APT-1008) Low Dose; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo Baseline vs EUR-1008 (APT-1008) High Dose; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Change From Placebo Baseline in Weight at End of Each Treatment Period
Description: Mean change from baseline in weight was calculated for end of treatment (6 days home treatment and 3-5 days hospital treatment) in first and second intervention periods.
Time Frame: Baseline, end of treatment (6 days home treatment and 3-5 days hospital treatment in first and second intervention periods)
Population: FAS included all participants who received at least one dose of the study medication. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | EUR-1008 (APT-1008) Low Dose | EUR-1008 (APT-1008) High Dose
Number analyzed (Participants) | 74 | 75
kilogram (kg) | 0.38 (1.18) | 0.50 (1.31)

5. Secondary Outcome: Change From Placebo Baseline in Body Mass Index (BMI) at End of Treatment
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2). Mean change from baseline in BMI was calculated for end of treatment (6 days home treatment and 3-5 days hospital treatment) in first and second intervention periods.
Time Frame: as for outcome 4
Population: FAS included all participants who received at least one dose of the study medication. Here "N" (number of participants analyzed) represents number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | EUR-1008 (APT-1008) Low Dose | EUR-1008 (APT-1008) High Dose
Number analyzed (Participants) | 74 | 75
kg/m^2 | 0.13 (0.39) | 0.16 (0.42)

ADVERSE EVENTS:
Time Frame: Baseline up to final follow-up visit (14 days after end of study)
Description: Adverse event (AE) was defined as any untoward medical occurrence regardless of causal relationship to study medication. Serious AE was any event that resulted in death, life threatening, required or prolonged in-patient hospitalization, significant disability/incapacity, or was a congenital anomaly/birth defect.
Groups:
- Placebo Baseline: Placebo matched to EUR-1008 (APT-1008) capsule orally daily for 4 days home treatment and 3 to 5 days hospital treatment in the baseline run-in phase, which were then randomized to either high dose or low dose of EUR-1008 (APT-1008).
Arm/Group | Placebo Baseline | EUR-1008 (APT-1008) Low Dose | EUR-1008 (APT-1008) High Dose
Serious Adverse Events (participants affected / at risk) | 2/82 | 2/74 | 2/75
Other Adverse Events (participants affected / at risk) | 34/82 | 28/74 | 31/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Baseline (N=82) | EUR-1008 (APT-1008) Low Dose (N=74) | EUR-1008 (APT-1008) High Dose (N=75)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Baseline (N=82) | EUR-1008 (APT-1008) Low Dose (N=74) | EUR-1008 (APT-1008) High Dose (N=75)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 7 | 13
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1
Flatulence (Gastrointestinal disorders) | 18 | 7 | 10
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 1
Steatorrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood glucose abnormal (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Blood uric acid decreased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 1 | 0
Protein induced by vitamin K absence or antagonist II increased (Investigations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin A deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin E deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 3 | 4 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus operation (Surgical and medical procedures) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with each agreement with the individual investigators. Sponsor will allow publication after a multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and can defer publication for a period of time to allow for Sponsor to obtain patent or other intellectual property right protection.